CLINICAL TRIAL: NCT05003648
Title: Treating Leg Symptoms in Women With X-linked Adrenoleukodystrophy: A Key to Improving Sleep and Gait Performance
Brief Title: Treating Leg Symptoms in Women With X-linked Adrenoleukodystrophy
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: European Leukodystrophy Association (Other)
Responsible Party: Principal Investigator, Florian Eichler, Associate Professor of Neurology, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021P001543
Record Dates: First submitted 2021-07-15; First posted 2021-08-12 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Adrenoleukodystrophy; Restless Legs Syndrome
MeSH Terms: conditions — Adrenoleukodystrophy; Restless Legs Syndrome | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will be on the placebo arm for 2 months and will then cross over to the pramipexole arm for 2 months
  Interventions: Drug: Placebo
- Pramipexole (Active Comparator): Participants will be on the pramipexole arm for 2 months and will then cross over to the placebo arm for 2 months
  Interventions: Drug: Pramipexole

INTERVENTIONS:
Drug: Pramipexole — Participants will be started on 0.125 mg pramipexole for the first week. If this dose is well tolerated but not effective, the dose can be increased to 0.25 mg for the following week. If this dose is well tolerated but not effective, the dose can be further increased to 0.5 mg for the remainder of the 2-month period.
  Arms: Pramipexole
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
The investigators recently observed that up to 25% of women with X-linked adrenoleukodystrophy (ALD) have moderate to severe Restless Leg Syndrome (RLS). In this study, the investigators aim to estimate the prevalence of RLS among women with ALD and to assess whether pramipexole improves RLS symptoms as well as sleep and gait measures in women with ALD.

DETAILED DESCRIPTION:
X-linked adrenoleukodystrophy (ALD) is a neurodegenerative disease caused by mutations in the ABCD1 peroxisomal half-transporter gene, resulting in accumulation of very long chain fatty acids (VLCFAs). As ALD is an X-linked disease, women were previously considered asymptomatic carriers. It is now known that even though adrenal insufficiency and cerebral disease occur in less than 1% of women, more than 80% eventually develop progressive spinal cord disease. Recently, the investigators observed that women are more frequently affected by movement disorders independent of the demyelinating brain disease seen in men. In a pilot study, the investigators found that up to 25% of women with ALD have moderate to severe Restless Leg Syndrome (RLS). RLS is a movement disorder characterized by a powerful urge to move the legs, usually accompanied by unpleasant dysesthesias, that is precipitated by rest, relieved by movement, and most pronounced in the evening or at night. Dopamine agonists such as pramipexole are efficacious and first-line FDA-approved treatments in low doses for primary (i.e., idiopathic) RLS and have been shown to improve both the primary symptoms of RLS (sensory discomfort, motor restlessness) as well as the associated sleep and quality of life impairments in RLS.

In the first phase of the study, the investigators will enroll 100 women with ALD at the two participating sites (Massachusetts General Hospital and University Medical Center Amsterdam). Participants will undergo structured phone interviews with both an expert in ALD and RLS to assess the presence of probable or definite RLS. Participants with probable or definite RLS will then undergo an additional phone call to determine RLS severity and assess eligibility for the second phase of the study. The objective of the first phase of the study is to determine the prevalence of RLS in women with ALD.

The second phase of the study will consist of a 4-month randomized, double-blind, placebo-controlled cross over study to assess whether pramipexole improves RLS symptoms as well as sleep and gait measures in women with ALD. The investigators will enroll 24 women with ALD and moderate to severe RLS. Participants will first be randomized 1:1 to 0.125-0.5 mg pramipexole or placebo. After the first two months, a switch-over visit will take place and include a battery of neurological assessments, walking measures, polysomnography, and questionnaires. At this visit, the crossover from pramipexole to placebo and from placebo to pramipexole will occur. The final study visit will occur 2 months after the switch-over visit and all study assessments will be repeated.

ELIGIBILITY:
PHASE 1 (PREVALENCE STUDY)

Inclusion Criteria:

1. Women of any ethnic origin.
2. Ability to provide verbal consent
3. A willingness and ability to comply with study procedures.
4. Age 18-75 years
5. Metabolically or genetically confirmed diagnosis of ALD

Exclusion Criteria:

1. Inflammatory brain demyelination

PHASE 2 (CROSS-OVER STUDY)

Inclusion Criteria:

1. Participation in Phase 1
2. Ability to provide written informed consent
3. Women with ALD who have Restless Leg Syndrome (IRLS > 15)

Exclusion Criteria:

1. Pregnant. Research staff perform pregnancy tests upon visit to center.
2. Participants with active or unstable major psychiatric disorder other than ALD, who, in the investigators' judgement, require further treatment
3. Use of dopaminergic agonists or antagonists within the last 30 days
4. Alcohol use disorder within the last 30 days
5. History of being treated for restless legs syndrome, specifically with dopamine agonist medications
6. Methamphetamine or benzodiazepine dependence in the last 30 days
7. Neurological disorder or cardiovascular disease raising safety concerns about use of pramipexole and/or judged to interfere with ability to assess efficacy of the treatment
8. Medical instability considered to interfere with study procedures
9. Renal disease judged to interfere with drug metabolism and excretion

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in the International Restless Legs Severity (IRLS) score | pre-intervention, week 8, week 17
  Change in IRLS score before and after pramipexole treatment. Scores range from 0 to 40, with higher scores representing more severe RLS symptoms.
Prevalence of Restless Leg Syndrome in Women with X-linked Adrenoleukodystrophy | pre-intervention
  The prevalence of RLS in women with ALD will be assessed using the Hening Telephone Diagnostic Interview (HTDI), an objective tool to diagnose RLS.

SECONDARY OUTCOMES:
Change in the 36-Item Short Form Survey (SF-36) score | pre-intervention, week 8, week 17
  Change in SF-36 score before and after pramipexole treatment. Scores range from 0 to 100, with higher scores representing better quality of life.
Change in the Generalized Anxiety Disorder Assessment (GAD-7) score | pre-intervention, week 8, week 17
  Change in GAD-7 score before and after pramipexole treatment. Scores range from 0 to 21, with higher scores representing more severe levels of anxiety.
Change in the Patient Health Questionnaire (PHQ-9) score | pre-intervention, week 8, week 17
  Change in the PHQ-9 score before and after pramipexole treatment. Scores range from 0 to 27, with higher scores representing more severe depression.
Improvement in RLS symptoms measured by the Clinical Global Impression - Improvement (CGI-I) scale | week 8 and week 17
  Improvement in the patient's illness after pramipexole treatment as determined by the physician. Scores range from 1 (very much improved) to 7 (very much worse).
Change in the Expanded Disability Status Scale (EDSS) score | pre-intervention, week 8, week 17
  Change in EDSS score before and after pramipexole treatment. Scores range from 0 (no disability) to 10 (death).
Change in the Multiple Sclerosis Walking Scale (MSWS-12) score | pre-intervention, week 8, week 17
  Change in MSWS-12 score before and after pramipexole treatment. Scores range from 0 to 100, with higher scores representing more severe walking impairment.
Change in the Suggested Immobilization Test (SIT) | pre-intervention, week 8, week 17
  Change in the sensory and motor aspects of RLS before and after pramipexole treatment, assessed using the SIT.
Change in sleep/wake parameters measured by actigraphy | pre-intervention, week 8, week 17
  Change in sleep/wake parameters including Total Sleep time, Sleep Latency, and Wake after Sleep Onset before and after pramipexole treatment. Parameters will be objectively measured using wrist-worn actigraphy.
Change in the Utah Early Neuropathy Scale (UENS) score | pre-intervention, week 8, week 17
  Change in UENS score before and after pramipexole treatment. Scores range from 0 to 42, with higher scores representing more severe neuropathy.
Change in the Timed Up and Go (TUG) Test | pre-intervention, week 8, week 17
  Change in the amount of time it takes for the patient to get up from an armchair, walk 3 m, turn around, walk back, and sit down again before and after pramipexole treatment. Higher scores represent more severe balance impairment.
Change in the 6 Minute Walk (6MW) Test | pre-intervention, week 8, week 17
  Change in the maximum distance a patient can walk in 6 minutes before and after pramipexole treatment. Higher scores represent better walking ability.
Change in quality of sleep and leg movements per hour of sleep measured by Polysomnography | pre-intervention, week 8, week 17
  Change in quality of sleep and indices of periodic leg movements before and after pramipexole treatment. These variables will be assessed using Polysomongraphy and will be measured at the Boston site only.
Change in the 13-item Spasticity Screening Tool score | pre-intervention, week 8, week 17
  Change in the Spasticity Screening Tool before and after pramipexole treatment. Scores range from 0 to 52, with higher scores representing more severe spasticity symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Florian S Eichler, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- University Medical Center of Amsterdam, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data will be shared between the two collaborating sites (Massachusetts General Hospital and University Medical Center of Amsterdam). We do not currently have a plan to share this data with other researchers.